CLINICAL TRIAL: NCT05317364
Title: Topical Vaginal Estrogen for Postpartum Obstetric Anal Sphincter Injury Recovery: a Randomized Clinical Trial
Brief Title: Topical Vaginal Estrogen for Postpartum Obstetric Anal Sphincter Injury Recovery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hannah Chapman, Clinical instructor, fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 300008970
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Obstetric; Injury Pelvic Floor; Sexual Dysfunction; Anal Incontinence; Urinary Incontinence
Keywords: Obstetric anal sphincter injury; sexual dysfunction; anal incontinence; urinary incontinence
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Encopresis; Urinary Incontinence | interventions — Estradiol; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive either topical vaginal estrogen or placebo cream and will continue this therapy for duration of study.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical vaginal estrogen group (Active Comparator): Estradiol vaginal cream 0.01% 1g will be administered vaginally, initiated at 2 weeks postpartum and continued until 6 months postpartum. Beginning at 2 weeks postpartum, 1g estradiol vaginal cream 0.01% will be administered by participants nightly for 2 weeks then twice weekly to complete 6 months therapy
  Interventions: Drug: Estradiol 0.01% Vag Cream
- Placebo group (Placebo Comparator): Placebo cream, 1g will be administered vaginally, initiated at 2 weeks postpartum and continued until 6 months postpartum. Beginning at 2 weeks postpartum, 1g of placebo cream will be administered by participants nightly for 2 weeks then twice weekly to complete 6 months therapy.
  Interventions: Drug: Placebo vaginal cream

INTERVENTIONS:
Drug: Estradiol 0.01% Vag Cream — 1g estradiol vaginal cream 0.01% or placebo will be administered nightly for 2 weeks then twice weekly to complete 6 months therapy
  Other Names: Estrace cream
  Arms: Topical vaginal estrogen group
Drug: Placebo vaginal cream — Placebo cream
  Other Names: Versabase vaginal cream
  Arms: Placebo group

SUMMARY:
Obstetric anal sphincter injuries (OASIS) cause significant morbidity and are well known risk factors for sexual dysfunction, urinary and anal incontinence. Postpartum and breastfeeding are relative hypoestrogenic states with risk factors for dyspareunia and vaginal atrophy. Estrogen deficiency results in changes in the vaginal epithelium and poor tissue quality which results in poor wound healing. For postmenopausal women with vaginal atrophy undergoing surgery for pelvic organ prolapse, early administration of topical vaginal E2 therapy resulted in improved markers of tissue quality. Currently, there are limited studies to reference for proposed treatment modalities to improve sexual function and incontinence in this population. In this proposed randomized, placebo-controlled trial, women who sustain OASIS will be recruited and randomized to begin intravaginal estrogen therapy or placebo at their 2-week follow-up visit after hospital discharge. Participants will complete validated questionnaires relating to sexual function and pelvic floor disorders (urinary and anal incontinence) symptom distress and impact. The primary outcome of this study will be sexual dysfunction symptom severity measured by the female sexual function index (FSFI) at 6 months postpartum. Secondary outcomes will be urinary and anal incontinence distress and impact measured by St. Mark's score and the fecal incontinence quality of life (FIQOL) questionnaire for anal incontinence and urogenital distress inventory (UDI-6) for urinary incontinence. The objective of this study is to determine if intra-vaginal estrogen therapy improves sexual function and incontinence symptom distress and impact for postpartum women after OASIS.

DETAILED DESCRIPTION:
Obstetric anal sphincter injuries (OASIS) are known to cause significant morbidity and are known risk factors for sexual dysfunction, urinary and anal incontinence. Recent studies have reported that women with OASIS experience more problems with sexual dysfunction compared to their age and parity matched counterparts who do not have these tears. Despite this, little attention is paid to its prevalence or treatment in this population. These women are also at a 4-fold higher risk of anal incontinence. Additionally, significantly more women with OASIS report urinary incontinence 10 weeks after delivery and have significantly worse quality of life scores. Postpartum and breastfeeding are relative hypoestrogenic states with risk factors for dyspareunia and vaginal atrophy. Estrogen deficiency results in changes in the vaginal epithelium and poor tissue quality which results in poor wound healing. For postmenopausal women with vaginal atrophy undergoing surgery for pelvic organ prolapse, early administration of topical vaginal E2 therapy resulted in improved markers of tissue quality.

Due to the significant morbidity associated with OASIS, it is critical to further explore treatment options to ultimately improve wound healing and outcomes in women who sustain OASIS tears in their postpartum recovery. Training in identification of OASIS and close follow up in specialized OASIS clinics have improved outcomes for these women. However, there are limited studies to reference for proposed treatment modalities to improve sexual function and incontinence in this population. Intra-vaginal estrogen therapy has proven to be safe and feasible in this population as demonstrated by no difference in the serum estrogen concentration in those women treated with intra-vaginal estrogen therapy for treatment of granulation tissue. Although evidence is limited, anecdotally, vaginal estrogen cream has been used to treat postpartum women with OASIS to treat vaginal atrophy and improve wound healing. This proposed research is critical to ultimately improving the postpartum recovery for women who sustain OASIS. This information will add to the growing literature aiming to optimize quality of life and improve care for these women.

In this proposed randomized, placebo-controlled trial, women who sustain OASIS will be recruited and randomized to begin intravaginal estrogen therapy or placebo at their 2-week follow-up visit, (upon establishing care at postpartum perineal clinic), after hospital discharge. Participants will complete validated questionnaires relating to sexual function and pelvic floor disorders (urinary and anal incontinence) symptom distress and impact at the 2-week postpartum visit (baseline). Participants will follow up at designated intervals (12-weeks and 6 months) and complete questionnaires with plan for total of 6-months intravaginal estrogen or placebo therapy. The primary outcome will be sexual dysfunction symptom severity measured by the female sexual function index (FSFI) at 6 months postpartum. Secondary outcomes will be urinary and anal incontinence distress and impact measured by St. Mark's and the fecal incontinence quality of life (FIQOL) scores for anal incontinence and urogenital distress inventory (UDI-6) for urinary incontinence. The objective of this study is to determine if intra-vaginal estrogen therapy improves sexual function and incontinence symptom distress and impact for postpartum women after OASIS. We hypothesize that topical vaginal estrogen cream therapy postpartum will improve sexual function scores thereby improving functional status and related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* women who sustained 3rd or 4th degree lacerations
* aged 18 years or older
* must be able to self apply vaginal cream

Exclusion Criteria:

* Contraindications to intra-vaginal estrogen therapy (spontaneous DVT, stroke, hormone responsive breast cancer)
* tobacco use
* allergy to estradiol vaginal cream 0.01% or its constitutions
* perineal wound breakdown or infection at 2-week Postpartum visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
sexual dysfunction symptom severity | 6 months postpartum
  measured by the female sexual function index (FSFI). Minimum score 1, maximum score 36. Higher scores indicate a higher level of sexual function.

SECONDARY OUTCOMES:
Urinary incontinence | 6 months postpartum
  measured by urogenital distress inventory (UDI-6). Minimum score is 0, maximum score 75. Higher scores indicate a higher level of distress and impact on quality of life caused by urinary incontinence.
Anal incontinence | 6 months postpartum
  measured by St. Mark's and the fecal incontinence quality of life (FIQOL) scores. For St. Marks, minimum score 0, maximum 24. A higher score indicates a higher degree of incontinence and impact on lifestyle. For FIQOL, minimum score is 4, maximum score is 20. A lower score indicates a lower functional status and related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah L Chapman, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sayed Ahmed WA, Kishk EA, Farhan RI, Khamees RE. Female sexual function following different degrees of perineal tears. Int Urogynecol J. 2017 Jun;28(6):917-921. doi: 10.1007/s00192-016-3210-6. Epub 2016 Dec 6. PMID 27924373
- [Background] Andrews V, Thakar R, Sultan AH, Jones PW. Evaluation of postpartum perineal pain and dyspareunia--a prospective study. Eur J Obstet Gynecol Reprod Biol. 2008 Apr;137(2):152-6. doi: 10.1016/j.ejogrb.2007.06.005. Epub 2007 Aug 2. PMID 17681663
- [Background] Soerensen MM, Buntzen S, Bek KM, Laurberg S. Complete obstetric anal sphincter tear and risk of long-term fecal incontinence: a cohort study. Dis Colon Rectum. 2013 Aug;56(8):992-1001. doi: 10.1097/DCR.0b013e318299c209. PMID 23838869
- [Background] Stedenfeldt M, Pirhonen J, Blix E, Wilsgaard T, Vonen B, Oian P. Anal incontinence, urinary incontinence and sexual problems in primiparous women - a comparison between women with episiotomy only and women with episiotomy and obstetric anal sphincter injury. BMC Womens Health. 2014 Dec 16;14:157. doi: 10.1186/s12905-014-0157-y. PMID 25511413
- [Background] Scheer I, Andrews V, Thakar R, Sultan AH. Urinary incontinence after obstetric anal sphincter injuries (OASIS)--is there a relationship? Int Urogynecol J Pelvic Floor Dysfunct. 2008 Feb;19(2):179-83. doi: 10.1007/s00192-007-0431-8. Epub 2007 Aug 2. PMID 17671753
- [Background] Woodward AP, Matthews CA. Outcomes of revision perineoplasty for persistent postpartum dyspareunia. Female Pelvic Med Reconstr Surg. 2010 Mar;16(2):135-9. doi: 10.1097/SPV.0b013e3181cc8702. PMID 22453161
- [Background] Karp DR, Jean-Michel M, Johnston Y, Suciu G, Aguilar VC, Davila GW. A randomized clinical trial of the impact of local estrogen on postoperative tissue quality after vaginal reconstructive surgery. Female Pelvic Med Reconstr Surg. 2012 Jul-Aug;18(4):211-5. doi: 10.1097/SPV.0b013e31825e6401. PMID 22777369
- [Background] Ripperda CM, Maldonado PA, Acevedo JF, Keller PW, Akgul Y, Shelton JM, Word RA. Vaginal estrogen: a dual-edged sword in postoperative healing of the vaginal wall. Menopause. 2017 Jul;24(7):838-849. doi: 10.1097/GME.0000000000000840. PMID 28169915
- [Background] Bochenska K, Kujawa S, Zhao H, Kenton K, Bulun SE, Lewicky-Gaupp C. Molecular Effects of Topical Estrogen on Vaginal Granulation Tissue in Postpartum Women. Female Pelvic Med Reconstr Surg. 2021 Aug 1;27(8):521-526. doi: 10.1097/SPV.0000000000001076. PMID 34261104
- [Background] Brown O, Heliker BD, Geynisman-Tan J, Tavathia M, Mueller MG, Collins S, Kenton K, Lewicky-Gaupp C. Vaginal Electrical Stimulation for Postpartum Neuromuscular Recovery: A Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Nov 1;27(11):659-666. doi: 10.1097/SPV.0000000000001037. PMID 34608032